CLINICAL TRIAL: NCT01251120
Title: A Pragmatic, Randomized, Parallel Group Study of the Effect on Disease Remission, Work Productivity and Tolerability of Tocilizumab in Combination With DMARDs and Individually Designed Best Practice DMARD Therapy in Patients With Early, Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Combination With DMARDs Versus Current Best Practice DMARD Therapy in Patients With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped prematurely due to lack of enrollment.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25346
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Antirheumatic Agents

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]
- 2 (Active Comparator)
  Interventions: Drug: DMARD

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg intravenously every 4 weeks plus background DMARDs (including methotrexate)
  Arms: 1
Drug: DMARD — Non-biologic DMARDs (including methotrexate) according to current best practice
  Arms: 2

SUMMARY:
This randomized, open-label, parallel-group study will assess the effect on disease remission of RoActemra/Actemra (tocilizumab) in combination with disease-modifying antirheumatic drugs (DMARDs) versus current best practice non-biologic DMARD therapy in patients with moderate-to-severe active rheumatoid arthritis. Patients who are randomly assigned to the RoActemra/Actemra treatment group will receive 8 mg/kg RoActemra/Actemra intravenously every 4 weeks. The anticipated time on study treatment is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, over the age of 18 years
* Diagnosis of moderate-to-severe active early rheumatoid arthritis (RA) of less than 2 years duration
* DAS28 >3.2
* Swollen joint count (SJC) >/=6 (66 joint count), and tender joint count (TJC) >/=6 (68 joint count)
* Patients who have received DMARDs (including methotrexate) for 3-7 months

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months after baseline
* Rheumatic autoimmune disease other than rheumatoid arthritis (secondary Sjögrens syndrome or nodulosis with RA is permitted)
* Functional class III or IV as defined by ACR Classification of Functional Status in Rheumatoid Arthritis
* Prior history of or current inflammatory joint disease other than RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Finland (6):
  - Hämeenlinna
  - Helsinki
  - Jyväskylä
  - Kuopio
  - Riihimäki
  - Rovaniemi

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) intravenously every 4 weeks along with background disease-modifying antirheumatic drugs (DMARDs) including methotrexate. All participants who received methotrexate also received at least 5 mg oral folic acid weekly.
- Non-biologic DMARDs: Participants received non-biologic DMARDs (including methotrexate) according to current best practice. All participants who received methotrexate also received at least 5 mg oral folic acid weekly.
Period: Overall Study
Arm/Group | Tocilizumab | Non-biologic DMARDs
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Due to limited number of participants (n=2) the study was prematurely terminated.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg intravenously every 4 weeks plus background DMARDs (including methotrexate)
- Placebo: Participants received Non-biologic DMARDs (including methotrexate) according to current best practice
- Total: Total of all reporting groups
Arm/Group | Tocilizumab | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (0.0) | 48.2 (0.0) | 55.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Disease Remission at Month 12 Assessed Using the Disease Activity Score Based on 28-Joint Count (DAS28)
Description: The DAS28 is a combined index for measuring disease activity in Rheumatoid Arthritis (RA). The index includes swollen and tender joint counts (SJC and TJC), acute phase response, and general health status. For this study Erythrocyte sedimentation Rate (ESR) was to be used to calculate DAS28 score. The DAS28, which uses a 28 joint count, is derived from the original DAS which includes a 44 swollen joint count. The DAS28 has been validated in RA. The index is calculated using the following formula:
  DAS28 equals (=) 0.56 times (×) square root of √(TJC) plus (+) 0.28 × √(SJC) + 0.70 × ln(ESR) + 0.014 × GH Where, TJC28 = tender joint count on 28 joints, SJC28 = swollen joint count on 28 joints, ln = natural log, ESR measured as millimeters per hour (mm/hr), and GH = general health, which is participant's global assessment of disease activity (100-mm Visual Analog Scale [VAS]). DAS28 less than/equal to (≤) 2.6 defined remission.
Time Frame: Month 12
Population: Because of the limited number (n) of participants (n=2), the study was terminated prematurely. No statistical analysis could be performed.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg intravenously every 4 weeks along with background DMARDs including methotrexate. All participants who received methotrexate also received at least 5 mg oral folic acid weekly.
Arm/Group | Tocilizumab | Non-biologic DMARDs
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Hours Absent From Work
Description: Work productivity measures include absence from work (participant reported and registries), permanent work disability (pension, participant reported and registries), presenteeism (Quantity and Quality instrument, QQ).
Time Frame: Baseline and 6 and 12 months
Population: Because of the limited number of participants (n=2), the study was terminated prematurely. No statistical analysis could be performed.
Arm/Group | Tocilizumab | Non-biologic DMARDs
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants Achieving Disease Remission at Month 6 Assessed Using DAS28
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes SJC and TJC, acute phase response, and general health status. For this study ESR was to be used to calculate DAS28 score. The DAS28, which uses a 28 joint count, is derived from the original DAS which includes a 44 swollen joint count. The DAS28 has been validated in RA. The index is calculated using the following formula:
  DAS28 = 0.56 × √(TJC) + 0.28 × √(SJC) + 0.70 × ln(ESR) + 0.014 × GH Where, TJC28 = tender joint count on 28 joints, SJC28 = swollen joint count on 28 joints, ln = natural log, ESR measured as millimeters per hour (mm/hr), and GH = general health, which is participant's global assessment of disease activity (100-mm VAS). DAS28 ≤ 2.6 defined remission.
Time Frame: Month 6
Population: as for outcome 2
Arm/Group | Tocilizumab | Non-biologic DMARDs
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants Achieving Responses According to American College of Rheumatology (ACR) Criteria
Description: The ACR definition of response includes tender and swollen joint counts, VAS scales for pain, participant and investigator global assessment of disease activity, participant-assessed disability using Health Assessment Questionnaire (HAQ) and acute phase response.
Time Frame: Months 6 and 12
Population: as for outcome 2
Arm/Group | Tocilizumab | Non-biologic DMARDs
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants Achieving Remission at Months 6 and 12 Assessed Using Clinical Activity Disease Index (CDAI)
Description: The CDAI is a purely clinical index to measure disease activity. The index includes swollen and tender joint counts, participant global assessment of disease activity, and evaluator global assessment of disease activity (EGA).
Time Frame: Months 6 and 12
Population: as for outcome 2
Arm/Group | Tocilizumab | Non-biologic DMARDs
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline to Months 6 and 12 in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT F) Scores
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participants fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). Clinically relevant improvement is defined as a ≥5-point change from Baseline.
Time Frame: Baseline and Months 6 and 12
Population: as for outcome 2
Arm/Group | Tocilizumab | Non-biologic DMARDs
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline to Months 6 and 12 in European Quality of Life-5D (EQ-5D) Score
Description: EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQoL Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline and Months 6 and 12
Population: as for outcome 2
Arm/Group | Tocilizumab | Non-biologic DMARDs
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline to Months 6 and 12 in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score
Description: HAQ-DI includes 20 questions concerning participant's activities of daily life, grouped in 8 scales of 2 to 3 questions for each activity. To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Overall score was computed as the sum of the domain scores and divided by the number of domains answered. Total possible score range was 0-3 where 0=without difficulties; 1= with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all.
Time Frame: Baseline and Months 6 and 12
Population: as for outcome 2
Arm/Group | Tocilizumab | Non-biologic DMARDs
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was terminated prematurely due to lack of enrollment. Adverse events were recorded from the date of screening until study termination.
Arm/Group | Tocilizumab | Non-biologic DMARDs
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=1) | Non-biologic DMARDs (N=1)
Gastointestinal Disorder (Gastrointestinal disorders) | 1 | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.